CLINICAL TRIAL: NCT02292056
Title: Medication Safety and Contraceptive Counseling for Reproductive Aged Women With Psychiatric Conditions
Acronym: MSRP
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of California, San Diego (Other)
Collaborators: MotherToBaby (Unknown)
Responsible Party: Principal Investigator, Sheila Mody, Faculty, University of California, San Diego
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 131088
Record Dates: First submitted 2014-11-12; First posted 2014-11-17 (Estimated); Last update posted 2014-11-17 (Estimated); Status verified 2014-11

CONDITIONS: Mental Disorders; Contraception; Chemical Teratogen Exposure
MeSH Terms: conditions — Mental Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Counseling Group (Experimental): Participation in the study will be completed in a single session and will involve a pre-counseling questionnaire, followed by a pre-counseling quiz, individualized counseling session, post-counseling quiz and post-counseling questionnaire.
  Interventions: Behavioral: 1-on-1 counseling

INTERVENTIONS:
Behavioral: 1-on-1 counseling — 1. Precounseling questionnaire collecting demographic information, contraception information, and reasons for choosing contraceptive method
  2. Precounseling quiz: assess baseline level of knowledge regarding medication safety and contraceptive option.
  3. Counseling: completed by MotherToBaby counselor about the safety of their medications for use in pregnancy.
  4. 10 minute video entitled "The Contraceptive Choice Project: Which Birth Control Method is Right for You?" by Washington University in St. Louis.
  5. Post-Counseling Quiz to assess whether specialized training impacted their understanding of medication safety and contraceptive options.
  6. Post-Counseling Questionnaire: assess contraceptive plans and satisfaction with counseling

SUMMARY:
There is currently limited research that addresses the unique medication safety and family planning needs among women of reproductive age with psychiatric conditions. The study will research the feasibility of a novel individualized 1-on-1 counseling session at the Gifford Clinic in the Department of Psychiatry at UCSD that will help women in this population better understand: 1) which of their medications are safe to use in pregnancy, 2) provide education regarding the importance of using contraception and which contraceptive choices are available to them, and 3) raise awareness of any drug-drug interactions that may exist between their medications and their chosen method of contraception. Patients will be given questionnaire to assess their contraceptive utilization. They will also be given a before and after quiz to allow for an objective measure of the patient's increase in knowledge regarding medication safety and contraceptive choices as a result of the investigators intervention.

DETAILED DESCRIPTION:
Nearly half of all pregnancies in the general population in 2006-2010 were unintended. In addition, data from the National Survey of Family Growth shows that in 2006-2010, only 62.2% of women aged 15-44 in the United States are using some form of contraception. These statistics inherently suggest a need for additional education in the general population regarding contraceptive options. It is unknown how these statistics for the general population apply to women with psychiatric conditions. In addition, reproductive age women with psychiatric diagnoses have several unique family planning considerations, some of which are outlined below:

TERATOGENICITY OF PSYCHIATRIC MEDICATIONS:

Some women with psychiatric conditions may be on medications that are not safe for use in pregnancy and therefore may require counseling on their highly effective contraceptive options. These women may also have other environmental exposures to alcohol, tobacco and illicit drugs, so this may be an additional need for counseling about risk to a potential pregnancy. Other women in this population may become pregnant and stop using their psychiatric medications because they are unaware that their medications are safe to use in pregnancy. The United States Food and Drug Administration uses the following categories to rate the safety of using various pharmaceutical agents in pregnancy: A, controlled studies in humans fail to demonstrate a risk to the fetus in pregnancy; B, no evidence of risk to fetus in animal studies but no controlled studies for use in pregnant women; C, animal studies demonstrate an adverse effect on the fetus, but no controlled studies in humans; D, positive evidence of risk to fetus in human studies; and X, agent contraindicated in pregnancy because risks to fetus clearly outweigh potential benefits. Most psychotropic drugs used to treat bipolar disorder are category C or D. For example, lithium, a commonly prescribed mood stabilizer used as a first-line treatment for bipolar disorder, is associated with an increased risk of congenital cardiac abnormalities and is FDA category D for use in pregnancy. Also, valproate and carbamazapine, which are commonly used as mood stabilizers, have been associated with neural tube defects in the fetus and thus are also FDA category D for use in pregnancy.

CONTRACEPTION:

Women in this population may also wish to delay or avoid pregnancy due to the current state of their psychiatric condition and thus should be encouraged to use effective contraception. It has been shown that women with psychiatric diagnoses may interrupt their use of contraception due a variety of factors including: drug-drug interactions with their psychiatric medication, psychiatric hospitalization, loss of personal control over their medication administration, and preconceived notions of how contraception may impact their psychiatric condition or vice versa. Long-acting reversible contraceptive options, such as intrauterine devices (IUDs), requiring no patient compliance to achieve maximal efficacy may therefore be particularly well-suited options for these women. For these reasons, there may be a role for focused counseling in this population regarding options for safe, effective and reversible forms of contraception.

DRUG-DRUG INTERACTIONS:

Some women with psychiatric conditions are on medications that interact with combined hormonal contraceptives and may benefit from specialized counseling regarding which contraceptive options are safe for them to use. In 2010, the Centers for Disease Control and Prevention (CDC) published the United States Medical Eligibility Criteria (USMEC) in an effort to improve contraceptive safety guidance. The USMEC includes guidance on contraceptive safety for specific medications, including those commonly used to treat psychiatric illness. For example, carbamazapine, oxcarbazapine, lamictal, and topiramate, which are commonly prescribed for mood stabilization, increase the clearance rate of oral contraceptives; thus patients receiving one of these treatments should consider switching to an alternative form of contraception. The USMEC continues to be updated and will likely prove to be a valuable resource to optimize contraceptive counseling for these women.

This multidisciplinary research project involves a unique collaboration between the MotherToBaby Project, Reproductive Medicine at UCSD and Psychiatry at UCSD to deliver individualized contraceptive and teratogen counseling to women with psychiatric conditions. MotherToBaby California, formerly known as the CTIS Pregnancy Health Information Line, in the Department of Pediatrics at UCSD is a community-based organization founded 27 years ago which has been continuously funded at UCSD to provide direct-to-consumer and direct-to-health care provider counseling free of charge on the risks or safety of medications, chemicals, recreational drugs and alcohol, infectious or chronic disease, and medical conditions in pregnancy. The goal of MotherToBaby is to provide individualized risk assessments and referrals for further assistance or diagnostic testing to pregnant or breastfeeding women in order to prevent birth defects that are related to prenatal or breastfeeding exposures.

The proposed study will serve to investigate the feasibility of a novel type of counseling service that may uncover and address unmet family planning needs of reproductive age women with psychiatric diagnoses. The proposed project also promotes the utilization of the relatively new evidence-based USMEC contraceptive guidance from the CDC which has been endorsed by the American Congress of Obstetricians & Gynecologists and American Academy of Family Physicians.

ELIGIBILITY:
Inclusion Criteria:

* Presenting for follow up psychiatric visit
* Ethnic Background: will include only english speaking participants (MotherToBaby counselors are only able to speak English)
* Level of Education: No limitation
* Health Status: at least one psychiatric condition for which they are taking medication
* Sexually active with Men

Exclusion Criteria:

* Planning to become pregnant
* Not sexually active with men
* History of hysterectomy, bilateral oophorectomy, or surgical sterilization
* Decisionally impaired - using post-consent instrument to assess decisional capacity. If a potential participant does not score 100% on post-consent instrument, then she will be excluded from participation.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2013-09; Primary Completion 2015-10 (Estimated); Study Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
Increase in Patient Knowledge | 1 year
  Assessed with score delta between Pre-counseling and Post-counseling Quizzes

SECONDARY OUTCOMES:
Contraceptive Plans | 1 year
  Captured in Post-Counseling questionnaire
Utilization of Contraception | 1 year
  Captured in Pre-Counseling questionnaire
Baseline Medication Safety Knowledge | 1 year
  Captured in Pre-Counseling questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Sheila Mody, MD MPH, Principal Investigator — UCSD Department of Reproductive Medicine
Locations (1):
- Gifford Clinic at UCSD Outpatient Psychiatry, San Diego, California, United States

REFERENCES:
- [Background] Trussell J, Wynn LL. Reducing unintended pregnancy in the United States. Contraception. 2008 Jan;77(1):1-5. doi: 10.1016/j.contraception.2007.09.001. Epub 2007 Dec 3. No abstract available. PMID 18082659
- [Background] Chandra A, Martinez GM, Mosher WD, Abma JC, Jones J. Fertility, family planning, and reproductive health of U.S. women: data from the 2002 National Survey of Family Growth. Vital Health Stat 23. 2005 Dec;(25):1-160. PMID 16532609
- [Background] Curtis V. Women are not the same as men: specific clinical issues for female patients with bipolar disorder. Bipolar Disord. 2005;7 Suppl 1:16-24. doi: 10.1111/j.1399-5618.2005.00190.x. PMID 15762865
- [Background] Guedes TG, Moura ER, Almeida PC. Particularities of family planning in women with mental disorders. Rev Lat Am Enfermagem. 2009 Sep-Oct;17(5):639-44. doi: 10.1590/s0104-11692009000500007. PMID 19967211
- [Background] CDC. U.S. medical eligibility criteria for contraceptive use, 2010: adapted from the World Health Organization medical eligibility criteria for contraceptive use, 4th edition. MMWR 2010;59 (No. RR-4)
- [Background] Crawford P. Interactions between antiepileptic drugs and hormonal contraception. CNS Drugs. 2002;16(4):263-72. doi: 10.2165/00023210-200216040-00005. PMID 11945109
- [Background] Committee opinion no. 505: understanding and using the U.S. Medical Eligibility Criteria For Contraceptive Use, 2010. Obstet Gynecol. 2011 Sep;118(3):754-760. doi: 10.1097/AOG.0b013e3182310cd3. PMID 21860318
- See also: "The Contraceptive Choice Project: Which Birth Control Method is Right for You?" by Washington University in St. Louis — http://www.youtube.com/watch?v=u9SHoy1C3tU